CLINICAL TRIAL: NCT07357194
Title: Barriers to Renal Rehabilitation Among Patients With Kidney Failure in Governmental Hospitals in Cairo: A Cross-Sectional Study
Brief Title: Renal Rehabilitation Among Patients With Kidney Failure
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Merna Mabrouk Labib keriakous, Barriers to Renal Rehabilitation among Patients with Kidney Failure in governmental hospitals in Cairo: A Cross-Sectional Study, Cairo University
Other Study IDs: Under request from Cairo Unive
Record Dates: First submitted 2026-01-13; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Renal Failure Acute Chronic
Keywords: Renal failure; Renal rehabilitation; Exercises; Renal dialysis
MeSH Terms: conditions — Renal Insufficiency; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with kidney failure doing dialysis

SUMMARY:
The primary purpose of this study is to identify and analyze the barriers to renal rehabilitation among patients diagnosed with kidney failure in Cairo

DETAILED DESCRIPTION:
This study is a cross-sectional design aimed at identifying the barriers to renal rehabilitation among patients diagnosed with kidney failure in governemtnal hospitals in Cairo.

The sample size for this study was determined using G*POWER statistical software (version 3.1.9.2; Franz Faul, Universitat Kiel, Germany) and was based on a previous study by (Bossola et al., 2014). which reported a prevalence of 38.1%. The required sample size calculated for this study is N=155, with calculations made using a significance level (α) of 0.05 and a statistical power of 80%. This sample size is deemed appropriate for achieving the study's objectives and ensuring statistically significant results.

155 patients suffering from kidney failure will participate in the study. They will be selected randomly from the different governmental hospitals centers in Cairo, Informed consent Freely and voluntarily consent to participate in this research study (Effect of pelvic floor down-training exercise on females with idiopathic overactive bladder) under the supervision and direction of the researcher/ Merna Mabrouk A thorough description of the study procedures has been explained to me, and I understand that I may withdraw my consent and discontinue participation in this study research at any time without prejudice to me.

ELIGIBILITY:
Inclusion Criteria:

Participants must have a confirmed diagnosis of kidney failure,

* Participants must be 18 years of age or older
* Participants must be willing and able to provide written informed consent (Appendix I).
* Participants must be receiving treatment at one of the nephrology clinics in Cairo that are involved in the study.

Exclusion Criteria:

Severe Cognitive Impairment or Psychiatric Disorders

* Recent Participation in Similar Studies
* Acute Medical Condition
* Inability to Communicate
* Pregnancy
* Non-residency in Cairo
* Non-compliance with Treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: * Participants must have a confirmed diagnosis of kidney failure,
  * Participants must be 18 years of age or older
  * Participants must be willing and able to provide written informed consent (Appendix I).
  * Participants must be receiving treatment at one of the nephrology clinics in Cairo that are involved in the study.
  Severe Cognitive Impairment or Psychiatric Disorders
  * Recent Participation in Similar Studies
  * Acute Medical Condition
  * Inability to Communicate
  * Pregnancy
  * Non-residency in Cairo
  * Non-compliance with Treatment
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2024-11-17 (Actual); Primary Completion 2025-01-30 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Dialysis patients' perception regarding exercise benefits and barriers Questionnaire (DPEBBS) | 20 minutes
  The perception of dialysis patients regarding exercise benefits and barriers will be measured using the DPEBBS

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Therapy, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided